CLINICAL TRIAL: NCT02647151
Title: Comparative Intraindividual Study, About the Efficacy and Safety of Treatment of Actinic Keratoses With Photodynamic Therapy Between Acid Methyl Aminolevulinate Cream and Aminolevulinic Gel
Brief Title: Efficacy and Safety of Treatment of Actinic Keratoses With Photodynamic Therapy Between MAL Cream and ALA Gel
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Instituto Valenciano de Oncología (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MALvsALA; 2015-002408-97 (EudraCT Number)
Record Dates: First submitted 2015-12-30; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Actinic Keratosis
Keywords: Acid Methyl Aminolevulinate (MAL); Aminolevulinic Gel (ALA) and Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- METHYLAMINOLEVULINATE HYDROCHLORIDE (Active Comparator): METHYLAMINOLEVULINATE HYDROCHLORIDE (MAL)cream 160mg/g. Intervention: Just one application of the product in the actinic keratosis lesions before the photodynamic therapy
  Interventions: Drug: METHYLAMINOLEVULINATE HYDROCHLORIDE; Drug: AMINOLEVULINIC ACID HYDROCHLORIDE
- AMINOLEVULINIC ACID HYDROCHLORIDE (Experimental): AMINOLEVULINIC ACID HYDROCHLORIDE (ALA) gel 78mg/g. Intervention: Just one application of the product in the actinic keratosis lesions before the photodynamic therapy
  Interventions: Drug: METHYLAMINOLEVULINATE HYDROCHLORIDE; Drug: AMINOLEVULINIC ACID HYDROCHLORIDE

INTERVENTIONS:
Drug: METHYLAMINOLEVULINATE HYDROCHLORIDE — This is an intrapatient randomized clinical trial. All patients participating in the trial will receive both, experimental and control treatment, randomization will be used to determine side (right or left for treatment). Three visits will be scheduled. In the first visit epidemiological data will be collected , Actinic Keratoses are counted and drawn in a transparent template and also a photograph of each side. In that first visit treatment the PDT will be also performed, the degree of fluorescence, the pain and the degree of immediate local reaction will be measured.
  skin after PDT. In the second visit, to be held at 2 or 3 days, the delayed local reaction degree will be assessed. And in the third visit, held a month of PDT the clinical response and patient satisfaction will be assessed.
  Other Names: MAL
Drug: AMINOLEVULINIC ACID HYDROCHLORIDE — This is an intrapatient randomized clinical trial. All patients participating in the trial will receive both, experimental and control treatment, randomization will be used to determine side (right or left for treatment). Three visits will be scheduled. In the first visit epidemiological data will be collected , Actinic Keratoses are counted and drawn in a transparent template and also a photograph of each side. In that first visit treatment the PDT will be also performed, the degree of fluorescence, the pain and the degree of immediate local reaction will be measured.
  skin after PDT. In the second visit, to be held at 2 or 3 days, the delayed local reaction degree will be assessed. And in the third visit, held a month of PDT the clinical response and patient satisfaction will be assessed.
  Other Names: ALA

SUMMARY:
Photodynamic therapy technique (PDT) is a conventional technique which is performed applying the product under occlusion lesions, let it incubate for 3 hours and then exposed skin to a light source, usually red.

The conclusions of efficacy, tolerance and satisfaction that today are known about PDT with MAL, but not with ALA, which is a new photosensitizer indicated for Actinic Keratoses. The pharmaceutical form of ALA is a gel, which gives a hypothetical better penetration and consequently it is more effectively.

DETAILED DESCRIPTION:
Intraindividual comparative study, to evaluate efficacy and safety of the treatment of actinic keratosis with photodynamic therapy between methyl aminolevulinate cream (MAL) and aminolevulinic acid nanosoma gel (ALA).

MAL cream: is an antineoplastic agent used as a photosensitizer for photodynamic therapy (PDT). The mode of action of methyl aminolevulinate in PDT was shown in the pharmacodynamic (PD) studies. In the target cells,methyl aminolevulinate was converted to photoactive porphyrins, including protoporphyrinIX (PpIX), which are the active photosensitizers. Upon light activation, the photosensitizers give rise to the production of cytotoxic singlet oxygen species which destroy the target cells.

ALA gel: Following topical application of 5-aminolaevulinic acid, the substance is metabolized to protoporphyrin IX, a photoactive compound which accumulates intracellularly in the treated actinic keratosis lesions. Protoporphyrin IX is activated by illumination with red light of a suitable wavelength and energy. In the presence of oxygen, reactive oxygen species are formed. The latter causes damage of cellular components and eventually destroys the target cells.

Photodynamic therapy technique (PDT) is a conventional technique which is performed applying the product under occlusion lesions, let it incubate for 3 hours and then exposed skin to a light source, usually red.

The conclusions of efficacy, tolerance and satisfaction that today are known about PDT with MAL, but not with ALA, which is a new photosensitizer indicated for QA. The pharmaceutical form of ALA is a gel, which gives a hypothetical better penetration and consequently it is more effectively.

ELIGIBILITY:
Inclusion Criteria:

1 Patient over 18 years old and capable of giving informed consent.

2. Provide at least 5 QA in two symmetrical areas of the face or scalp.

3. Accept the abandonment of sun creams and other creams (retinoic hydroxy acids, emollients, Topical Antibiotics ) in the treatment area during the time of the study.

4. Accept that it will postpone the treatment of other actinic keratosis close to treatment area.

5. Accept to go to scheduled visits. They should answer a questionnaire about epidemiology, history and treatment satisfaction. They will accept a photo of treatment area at each visit.

Exclusion Criteria:

1. Have any dermatological disease on the treatment zone or around it.
2. Patients who have previously been treated with therapy Photodynamic in targeted areas.
3. Patients with alcohol or drug dependence.
4. Patients who are currently participating in other studies.
5. Patients who have received any of the following medications at a time less than the indicated:

   * Systemic chemotherapy in the last 6 months.
   * Retinoids systemic , interferon , immunomodulatory or immunosuppressive , cytotoxic including agents , corticosteroids systemic , in the last month .
   * Ultraviolet A light, Ultraviolet B light, ablative laser, dermabrasion, chemical peels, in the last 6 months.
   * Topical retinoids , topical 5 -fluorouracil in the last month.
   * Cryotherapy , surgical excision, curettage, topical corticosteroids in the last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of MAL with the new BF -200 ALA photosensitizer in actinic keratosis. The Immediate and Delayed Local Reaction and Tolerance will be measured to compare MAL and ALA. | 1 month
  The main objective of this study is to compare the MAL with the new BF -200 ALA photosensitizer in terms of local reaction and tolerance for the treatment of actinic keratosis .
  First of all, the immediate local reaction to the lighting may include a greater or less erythema, inflammation and edema. It is scored on a scale of 0-10 where 0 is normal skin without local reaction and 10 is a maximum local reaction.
  The delayed local reaction is defined by the presence in different degrees of erythema, swelling, edema, pustules and scabs. They are also marked from 0 to 10 where 0 is normal skin without reaction and 10 for local maximum reaction.
  On the other hand, tolerance will be measured by the number, frequency and grade of reported adverse events in patients.

SECONDARY OUTCOMES:
Comparison of the clinical response measured by the efficacy and characteristics of fluorescence emission between the two photosensitizers. Partial and total response will be defined with ≥75% (partial response) and 100% (complete response.) | 1 month
  To compare the efficacy and characteristics of fluorescence emission between the two photosensitizers.
  The efficacy will be assessed by the initial photography and the template transparent. Both of them are measured at the beginning of the study and at the end of the study.
  Partial response will be defined if ≥75% of initial response of Actinic Keratosis is solved and complete response (CR) lf 100% of Actinic Keratosis is solved.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Serra, Principal Investigator — Servicio Dermatologia FIVO
Locations (1):
- Fundación instituto valenciano de Oncología, Valencia, Valencia, Spain